CLINICAL TRIAL: NCT05542719
Title: Mexican Registry of Dyslipidemia in Patients at High and Very High Risk of Atherosclerotic Cardiovascular Disease and the Use of an Application to Achieve Dyslipidemic Treatment Goals - REMEXDIS-IMSS
Brief Title: Mexican Registry of Dyslipidemia in Patients at High Risk and Very High Risk of Atherosclerotic Cardiovascular
Acronym: REMEXDIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Martha Alicia Hernandez Gonzalez, Head of health research division Centro Medico Nacional Bajio Umae T1 Leon Guanajuato, Coordinación de Investigación en Salud, Mexico
Other Study IDs: R-2021-785-103
Record Dates: First submitted 2022-09-08; First posted 2022-09-15 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Secondary Prevention; Cardiovascular Disease With Mention of Arteriosclerosis; Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- frequency of dyslipidemias: To describe the frequency of dyslipidemias in high-risk and very high-risk patients with atherosclerotic cardiovascular disease and analyze the impact of using an application to achieve dyslipidemia treatment goals at one-year follow-up.
  Interventions: Other: application

INTERVENTIONS:
Other: application — Through the application, determine if the patient is out of LDL-C goals for referral and treatment review.
  Show the usefulness of the application in achieving dyslipidemia treatment goals in patients with high and extremely high cardiovascular risk

SUMMARY:
Background. Atherosclerotic cardiovascular disease (ACVD) comprising coronary disease, cerebrovascular disease, peripheral artery disease, and aortic atherosclerosis caused 8.9 million deaths worldwide according to reports submitted by the World Health Organization during 2019, the development and progression of atherosclerosis is favored in the presence of modifiable risk factors such as dyslipidemia. In Mexico, during the period from December 29, 2019, to August 29, 2020, 141,873 deaths from heart disease were reported, even above the 108,658 deaths from SARS COV2 in the same time period. Although it is known that the Mexican mestizo population is susceptible to certain metabolic lipid disorders related to genetic variants, the frequency of dyslipidemia in patients with high cardiovascular risk is unknown to date and may be responsible for this increase. On the other hand, it has been shown that lowering LDL-C levels in this population by means of the pharmacological or dietary treatment stated the current guidelines, decreases chance of death, heart failure, angina, re-infarction or need for coronary revascularization; however, there are still patients not achieving treatment goals. Consequently, it is suggested that through the implementation and correct use of technological tools it is possible to increase efficiency in the medical follow-up of patients, allowing for appropriate lipid levels, like other chronic degenerative diseases such as diabetes and systemic arterial hypertension.

Objective. To describe the frequency of dyslipidemias in high-risk and very high-risk patients with atherosclerotic cardiovascular disease, who are IMSS beneficiaries, and to analyze the impact of using an application to achieve dyslipidemia treatment goals at one-year follow-up. Hypothesis For the National Register: Not required since the main objective is to carry out a national register of dyslipidemias. For the use of the application: Null hypothesis: The use of the application does not change the frequency of patients with high and extremely high atherosclerotic cardiovascular risk who achieve the goals of dyslipidemia treatment during one year of follow-up.

DETAILED DESCRIPTION:
Material and Methods. Design and selection criteria. This is a cuasi experimental with temporal series measures, multicenter, in adult patients entitled to the IMSS who are treated in different hospitals of the three levels of care, meeting the definition of elevated risk or extremely elevated risk of atherosclerotic cardiovascular disease. Those who lose validity, pregnant or nursing women, or who do not want to continue participating in the study will be excluded. Patients with acute coronary ischemic syndrome should wait two months to be included in the study. Sample size. Calculation of sample size was estimated according to the ODISSEY study, where the frequency of the cardiovascular event or outcome was 11.3% for those receiving the maximum treatment and therefore with adequate lipid levels, and 9.8% for those that do not, assuming a significance level of 0.05, 17,116 registered patients, with initial evaluations, and at 1, 3, 6, and 12 months. Methods. Clinical and laboratory measurements will be made at each appointment and the data will be uploaded to dedicated loaded database. The Portable Test Strip Analyzer (CardioChek) shall be used for glucose and lipid profile measurement and if the treatment target has not been achieved (LDL-C < 70 mg/dL or < 1.8 mmol/L), the application will issue an alert to the health personnel involved for their knowledge, and to be attended in a timely and priority manner at the specialty consultation assigned to them, and an alert will be sent to the patient, reminding them their next appointment.

Variables. Grouping: High-risk patients and extremely high cardiovascular risk. Primary. Dyslipidemia/Dyslipidemia Treatment Goal with the use of the applicative. The goal to achieve is to maintain an LDL-C value <70 mg/dL or <1.8 mmol/L.Secondary. Age, gender, diabetes mellitus, hypertension, obesity, weight, height, schooling, and treatment used. Explorative: Cardiac and non-cardiac mortality, unstable angina requiring hospitalization, non-fatal myocardial infarction, fatal or non-fatal ischemic cerebral vascular disease, need for surgical or percutaneous coronary revascularization. Lipid-lowering treatment used.

Statistical management of information. Exploratory analysis. The type of distribution of the continuous quantitative variables shall be determined according to the bias and kurtosis values and the Kolmogorov-Smirnov test shall establish whether they have normal distribution or not.

Descriptive analysis. Qualitative variables such as biological sex and presence of major cardiovascular event shall be expressed as frequency or proportion and continuous quantitative variables such as age and lipid levels as mean and standard deviation if they follow normal distribution or as median and percentiles otherwise.

Inferential analysis. For the National Register. The investigators will identify if there are differences between patients with extremely elevated risk and elevated risk for qualitative variables such as biological sex, schooling, treatment used, absolute number of risk factors, etc., by means of chi square test (or Fisher exact as the case may be) and risk will be calculated by odds ratio with their respective confidence interval. To identify whether there are differences between groups of quantitative variables such as systemic arterial pressure, waist circumference, lipid levels, etc., the comparison will be performed by Student's t-test for independent variables (or Mann Whitney U if the data do not have normal distribution). A logistic regression analysis will be performed to identify the weight of each variable in relation to the risk classification, this being the regressor to be included in the model.

For the use of the application. The investigators will analyze the proportion of patients who reached the treatment goal, identify when the highest proportion of patients reach the therapeutic goal, and whether there is variation in the proportion of patients who achieve the treatment goal at different timepoints by means of the square xi test. To identify the presence of major cardiovascular events, during follow-up, event freedom curves were performed, comparing the very high risk and high risk levels according to whether they achieved the treatment goal - LDL-C at <70 mg/dL or <1.8 mmol/L, Mantel Cox's proportional risk analysis will also be performed, and the weight of each variable will be identified with logistic regression in the outcome variables, these being the regressors that will be included in the model.

All information will be recorded in an ex profeso database and for all inferential statistical analyzes, significant p-values less than 5% will be considered. MedCalc v. statistical packages 20.1 and/or SPSS 20 will be used for analysis.

The statistical analysis will be performed by the expert statistician involved in the project.

ELIGIBILITY:
Inclusion Criteria:

* Adults, over 18 years old, Both biological sexes, And having any of the following characteristics

  1. Recurring atherosclerotic disease (2 or more events of atherosclerotic cardiovascular disease)
  2. Atherosclerotic cardiovascular disease plus

     * type 1 or type 2 diabetes mellitus with over 20 years of evolution,
     * Chronic renal failure with glomerular filtration rate lower than 30 mL/min or receiving dialysis or hemodialysis.
     * History of familial hypercholesterolemia in 1° or 2° degree.
  3. At least one of the following factors

     * Cholesterol ≥310 mg/dL (8 mmol/L) and/or LDL-C ≥190mg/dL and/or blood pressure ≥180/110 mmHg.
     * Familial hypercholesterolemia at 1° or 2° without other risk factors.
     * Diabetes mellitus without damage to target organ or more than 10 years of evolution plus another risk factor such as hypertension, dyslipidemia, or active smoking
     * Chronic renal failure with glomerular filtration between 30 and 59 mL/min.

Exclusion Criteria:

* Patients with acute coronary syndrome in the last two months
* Patients requiring hospitalization.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who attend outpatient service of family medicine, internal medicine, cardiology, or endocrinology of hospitals of first, second or third level of care of the Mexican Institute of Social Security and who meet the definition of elevated risk or extremely elevated risk of atherosclerotic cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 13166 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
National Register | 1 year
  Frequency of dyslipidemia according to the geographic region of the country.
use of the application | 2 years
  Usefulness of the application in achieving dyslipidemia treatment goals in patients with high and extremely high cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Martha A Hernandez, Gonzalez, Principal Investigator — CIS Mexico; Juan P Fernandez, Hernandez, Principal Investigator — CIS Mexico
Locations (1):
- Umae Cmn T1, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided